CLINICAL TRIAL: NCT02803125
Title: Improving Psychosocial Functioning in Older Veterans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D1832-W
Record Dates: First submitted 2016-05-19; First posted 2016-06-16 (Estimated); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; Aging; Veteran; Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Developed psychosocial intervention (Active Comparator): The active intervention in this study that will be compared to support group control
  Interventions: Behavioral: Psychosocial intervention
- Support group control (Placebo Comparator): This is the comparison group
  Interventions: Behavioral: Support group control

INTERVENTIONS:
Behavioral: Psychosocial intervention — This intervention is to be developed during the study. It will likely include modules that provide anger management strategies, communication skills, and education about interpersonal relationships and social support. In addition, psychoeducation about behavioral activation and stress management will likely be included
  Arms: Developed psychosocial intervention
Behavioral: Support group control — The support groups will be process-oriented in nature with core elements manualized to facilitate consistency of the intervention. In particular, group leaders will facilitate a check-in with the group, and the agenda will be open to topics brought in by group members
  Arms: Support group control

SUMMARY:
The purpose of this project is to develop an intervention to improve psychosocial functioning and quality of life for older Veterans with partial or full PTSD.

DETAILED DESCRIPTION:
This project will develop, implement, and evaluate a group protocol geared toward restoring older Veterans to better, fuller functioning. This project will determine the feasibility and acceptability of such an intervention. The intervention developed will then be compared to a support group control condition. Primary outcomes are psychosocial functioning and quality of life, with PTSD and depressive symptoms as secondary outcomes. A complementary objective is to improve attitudes toward mental health treatment and to increase readiness for change and engagement in evidence-based psychotherapies, as appropriate. Results from this study will provide feasibility data for future development and testing of the intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

Focus groups:

* Veterans need to be at least 60 years old to be eligible to participate in the focus groups.
* Potential participants will be assessed with the Primary Care Posttraumatic Stress Disorder Screener (PC-PTSD-5) prior to being invited to participate.
* Inclusion criteria include endorsement of a military-related criterion A event and a score of 3 or higher on the PC-PTSD-5.

Pilot:

* Veterans need to be at least 60 years old to be eligible to participate in the study.
* Potential participants will be assessed for PTSD symptoms.
* Inclusion criteria include endorsement of a military-related criterion A event and several PTSD symptoms.

Comparison:

* Veterans need to be at least 60 years old to be eligible to participate in the study.
* For both intervention and support groups, participants (who will be assessed for PTSD), must endorse a military-related criterion A event and several PTSD symptoms.

Exclusion Criteria:

Focus groups:

* Veterans who are diagnosed with a psychotic disorder or have psychotic symptoms, have been hospitalized for suicidal ideation or psychosis within the past year, or have a diagnosis of dementia or other severe cognitive disorder.
* Potential participants will also be excluded if they do not agree to be audio recorded.

Pilot:

* Veterans who are in current treatment for PTSD, are diagnosed with a psychotic disorder or have psychotic symptoms, have been hospitalized for suicidal ideation or psychosis within the past year, or have a diagnosis of dementia or other severe cognitive disorder.
* Veterans will be asked not to join therapy groups or other interventions for the duration of their participation in the study.
* Potential participants will also be excluded if they do not agree to be audio recorded.

Comparison:

* Veterans who are in current treatment for PTSD, are diagnosed with a psychotic disorder or have psychotic symptoms, have been hospitalized for suicidal ideation or psychosis within the past year, or have a diagnosis of dementia or other severe cognitive disorder.
* Veterans will be asked not to join therapy groups or other interventions for the duration of their participation in the study.
* Potential participants will also be excluded if they do not agree to be audio recorded.
* In addition, Veterans who participated in the pilot phase of the study will be excluded from participating in the comparison condition phase.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anica Pless Kaiser, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Any data to be shared will be coded data within a limited dataset, with appropriate Data Use Agreement (DUA) in place.

REFERENCES:
- [Derived] Pless Kaiser A, Ream M, Spiro A, Sloan DM, Cook JM, Vogt D, Moye JA. Feasibility, acceptability, and outcomes: A pilot trial of the enhancing social function in older veterans with PTSD (ESVP) group intervention. Psychol Serv. 2025 Jun 26:10.1037/ser0000962. doi: 10.1037/ser0000962. Online ahead of print. PMID 40569724
- [Derived] Pless Kaiser A, Daks JS, Korsun L, Heintz H, Moye J, Sloan DM, Cook JM, Vogt D, Spiro A 3rd. Enhancing social functioning in older veterans with PTSD: Rationale and design of an intervention and initial RCT. Contemp Clin Trials. 2024 Apr;139:107485. doi: 10.1016/j.cct.2024.107485. Epub 2024 Mar 2. PMID 38432471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Developed Psychosocial Intervention | Support Group Control
Started | 18 | 16
Completed | 13 | 12
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Developed Psychosocial Intervention | Support Group Control | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.56 (5.56) | 73.56 (4.41) | 71.97 (5.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 14 | 15 | 29
  Race/Ethnicity: Black or African American | 3 | 1 | 4
  Race/Ethnicity: Unanswered | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 16 | 34
Inventory of Psychosocial Functioning - Romantic [Mean (Standard Deviation); unit: units on a scale] — Lower scores indicate less impairment; Range = 0 - 66.
  units on a scale | 27.5 (11.0) | 17.0 (12.3) | 24.34 (11.84)
Quality of Life Inventory [Mean (Standard Deviation); unit: T-score] — Higher scores indicate greater quality of life; T scores values (e.g., range 0 - 100, 50 indicates the population mean with a standard deviation of 10).
  T-score | 32.83 (2.58) | 34.38 (2.63) | 33.48 (2.69)
VR-12 [Mean (Standard Deviation); unit: T-score] — T-scores (e.g., range 0 - 100, 50 indicates the population mean with a standard deviation of 10); Higher scores indicate better functioning
  T-score
    Mental Health Summary | 41.31 (8.85) | 42.36 (7.96) | 41.75 (8.37)
    Physical Health Summary | 39.01 (8.27) | 35.04 (10.78) | 37.34 (9.45)

OUTCOME MEASURES:

1. Primary Outcome: Inventory of Psychosocial Functioning (IPF) - Romantic, Family, Friends/Socializing Subscales
Description: The IPF is an 80-item self-report measure designed to assess functional impairment experienced by Veterans. Respondents rate how often they have acted a certain way over the past 30 days. Items are rated on a 7-point scale ranging from 0 ("never") to 6 ("always"). The IPF yields a total score (0-66) and scores for seven subscales: romantic relationships, family, work, friendships and socializing, parenting, education, and self-care functioning (lower indicates better functioning/less impairment). Respondents have the option to skip sections that do not apply to them. The IPF has excellent internal consistency reliability (overall alpha = .93) and the scale correlates with other self-report measures of quality of life and functional impairment, such as the QOLI (r = .59). Reporting on romantic relationships (range = 0-66), family (range = 0-42), and friends/socializing (range = 0-48) functioning subscales here. Higher scores indicate more impairment.
Time Frame: Reporting on baseline and post-group assessment (assessed at the final group session, approximately 2.5 - 3 months after baseline)
Population: Veterans who completed baseline and post-group assessments (assessed at the final group session). The number analyzed is different from the number who completed the study because not all participants completed enough items of each measure to be included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Developed Psychosocial Intervention | Support Group Control
Number analyzed (Participants) | 7 | 3
units on a scale
  IPF - romantic | 24.1 (10.0) | 15.7 (4.0)
  IPF - Family | 12.2 (9.9) | 17.5 (7.7)
  IPF - Friends/Social | 12.5 (6.4) | 15.4 (5.2)

2. Primary Outcome: Quality of Life Inventory (QOLI)
Description: The QOLI is a 32 item self-report measure that assesses life satisfaction across 16 life domains (e.g., health, work, recreation). For each domain, the respondent rates how important the domain is on a 0-2 scale and how satisfied he or she is in this area of life on a 7-point scale. Satisfaction scores on the measure are weighted based on the respondent's rating of the importance of the life domain in order to achieve a total score with higher scores indicating higher quality of life. The measure was validated across a number of samples, including psychiatric inpatient and outpatient VA samples. Test-retest reliability was excellent over a one-month interval (r = .91) as was the internal consistency of the measure (alphas ranged from .86-.89). The measure also demonstrated convergent and discriminant validity with other measures of life satisfaction. T scores were used with range 0 - 100, Mean (of reference population) =50, Standard deviation = 10
Time Frame: Reporting on baseline and post-group scores (assessed at the final group session, approximately 2.5 - 3 months after baseline)
Population: Baseline and post-group assessments (assessed at the last session of the intervention). The number analyzed is different from the number who completed the study because not all participants completed enough items of each measure to be included in the analysis.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Developed Psychosocial Intervention | Support Group Control
Number analyzed (Participants) | 13 | 10
T-scores | 34.69 (2.63) | 33.6 (1.90)

3. Primary Outcome: Veterans Rand 12-item (VR-12) Health Survey
Description: The VR-12 is a 12-item scale that assesses the effects of physical and mental health on well-being, and is often used to assess quality of life. Item scores are used to compute two broad component scores: the physical component score (PCS) and the mental component score (MCS). The component scores are standardized T-Scores and the population standard for this measure was recently updated. Higher scores indicate better functioning. T scores were used with range 0 - 100, Mean (of reference population) = 50, Standard deviation = 10
Time Frame: as for outcome 2
Population: Baseline and post-group scores (assessed at the final group session, approximately 2.5 - 3 months after baseline). The number analyzed is different from the number who completed the study because not all participants completed enough items of each measure to be included in the analysis.
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Developed Psychosocial Intervention | Support Group Control
Number analyzed (Participants) | 13 | 10
T-scores
  Mental Health Summary | 44.59 (9.55) | 40.37 (9.14)
  Physical Health Summary | 42.08 (8.15) | 37.44 (9.34)

ADVERSE EVENTS:
Time Frame: Data to inform adverse event reporting were collected during the entire data collection process that included participants. Monitoring/assessment for adverse events for each participant was completed through study completion, an average of about 8-9 months per participant.
Arm/Group | Developed Psychosocial Intervention | Support Group Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT02803125/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/25/NCT02803125/ICF_001.pdf